CLINICAL TRIAL: NCT03566849
Title: Effects of the Kinetic Chain Management Approach on Pain and Performance in Volleyball Athletes With Scapular Dyskinesia: A Randomized Controlled Trial
Brief Title: Effects of the Kinetic Chain Approach for Scapular Dyskinesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yi-Fen Shih, Professor, Department of Physical Therapy and Assistive Technology, National Yang-Ming University, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YM106028F
Record Dates: First submitted 2017-09-15; First posted 2018-06-25 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Volleyball; Shoulder impingement; Scapular dyskinesis; Kinetic chain
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial (RCT) with two treatment groups, kinetic chain management approach (KC) and conventional training of scapula dyskinesis (CT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KC group (Experimental): It mainly involve all segment in kinetic chain, not only shoulder girdle, include exercise training 3 times a week for a total 4 weeks.
  Interventions: Other: KC group
- CT group (Experimental): It involve shoulder girdle only, include exercise training 3 times a week for a total 4 weeks.
  Interventions: Other: CT group

INTERVENTIONS:
Other: KC group — 1. 1st week: each 10 rep/set, 3 set/day. PNF scapular pattern: posterior depression (Combination of isotonic, COI), Ball modified prone Cobra, Ball prone V-raise, Ball prone row, Ball side plank, Ball one-leg bridging
  2. 2nd week: each 10 rep/set, 3 set/day. Half sit-up with rotation to left/right, Side plank with ER, Prone extension with rotation to left/right, Bilateral one-leg squat with flexion, Squat to row
  3. 3rd week: 5 rep/set, 3 set/day (sling exercise). Prone shoulder protraction, Supine shoulder retraction, Side-lying hip ABD/ADD, Supine pelvic lift, Prone bridging
  4. 4th week: each 10 rep/set, 3 set/day. Lateral lunges with shoulder ABD/ER, Lunge with trunk rotation, Forward punch plus with serape effect, Spiking exercise, One-quarter vertical squat jump
  Other Names: Exercise therapy
  Arms: KC group
Other: CT group — 1. 1st week: each 10 rep/set, 3 set/day. PNF scapular pattern: posterior depression (Combination of isotonic, COI), Knee push up plus, Modified prone Cobra, Prone V-raise, Prone row, Side-lying ER
  2. 2nd week: each 10 rep/set, 3 set/day. Supine punch, Prone horizontal ABD, Prone V-raise, Prone row, Side-lying ER
  3. 3rd week: each 10 rep/set, 3 set/day. Sitting chest press, Sitting ABD in scaption, Sitting overhead press, Long-sitting resisted extension, Sitting ER
  4. 4th week: each 10 rep/set, 3 set/day. Standing horizontal pull-apart, Standing retraction plus ER, Standing resisted extension, Ball pushed on wall and controlled rolling, Wall push-up
  Other Names: Exercise therapy
  Arms: CT group

SUMMARY:
Volleyball is a highly technical sport which involved powerful overhead movements performed repetitively. Shoulder injuries is the third-most commonly injured body part in volleyball, with the majority resulting from chronic overuse. Abnormal scapular motions and positions relative to the thorax have been linked to various shoulder pathologies, including subacromial impingement, rotator cuff tears, and glenohumeral inferior instability. Also, Muscular imbalances around the shoulder complex could lead to dyskinesis and resulting in shoulder joint injuries (e.g. instability and impingement).

The concept of "kinetic chain" is coordinated sequencing of the segments. Sequential activation of the LE, pelvis and trunk muscles is required to facilitate the forces to be transferred appropriately from these body segments to the UE.

Reeser et al. have identified risk factors for volleyball-related shoulder pain and dysfunction. They found volleyball athletes who demonstrated core instability would show greater relevance to SICK scapula, and they also more likely to report a history of shoulder problems. Sciascia et al. also have reviewed that 49% athletes with posterior-superior labral tears showed either decreased hip rotators ﬂexibility or decreased hip abductors strength. Consequently, the deficits in kinetic chain segments would resulted in scapula dyskinesis, even lead to shoulder girdle dysfunction or injury.

Therefore, the modern training programs for athletes, especially in overhead players, should combine kinetic chain exercises to improve upper- and lower body core strength, sport-speciﬁc strength, performance, and prevent injury occurrence or recurrence.

In consideration of no randomized controlled trials (RCTs) have been performed to determine whether kinetic chain exercise would be more effective to conventional scapula training for patients with secondary shoulder impingement. The purpose of the study is to investigate the effects of kinetic chain management approach (KC) and conventional training of scapula dyskinesis (CT) in volleyball athletes with scapular dyskinesia. The investigators hypothesized that KC group would be more effective in self-reported pain, and their scapula would become more stable during movement task (arm-lifting and spiking) after a 4-week training program than CT group.

DETAILED DESCRIPTION:
Volleyball is a highly technical sport which involved powerful overhead movements performed repetitively. Shoulder injuries is the third-most commonly injured body part in volleyball, with the majority resulting from chronic overuse. Abnormal scapular motions and positions relative to the thorax have been linked to various shoulder pathologies, including subacromial impingement, rotator cuff tears, and glenohumeral inferior instability. Also, Muscular imbalances around the shoulder complex could lead to dyskinesis and resulting in shoulder joint injuries (e.g. instability and impingement).

The concept of "kinetic chain" is coordinated sequencing of the segments. Sequential activation of the LE, pelvis and trunk muscles is required to facilitate the forces to be transferred appropriately from these body segments to the UE.

One previous study have identified risk factors for volleyball-related shoulder pain and dysfunction. They found volleyball athletes who demonstrated core instability would show greater relevance to SICK scapula, and they also more likely to report a history of shoulder problems. Another study also have reviewed that 49% athletes with posterior-superior labral tears showed either decreased hip rotators ﬂexibility or decreased hip abductors strength. Consequently, the deficits in kinetic chain segments would resulted in scapula dyskinesis, even lead to shoulder girdle dysfunction or injury.

Therefore, the modern training programs for athletes, especially in overhead players, should combine kinetic chain exercises to improve upper- and lower body core strength, sport-speciﬁc strength, performance, and prevent injury occurrence or recurrence.

In consideration of no randomized controlled trials (RCTs) have been performed to determine whether kinetic chain exercise would be more effective to conventional scapula training for patients with secondary shoulder impingement. The purpose of the study is to investigate the effects of kinetic chain management approach (KC) and conventional training of scapula dyskinesis (CT) in volleyball athletes with scapular dyskinesia. The investigators hypothesized that KC group would be more effective in self-reported pain, and their scapula would become more stable during movement task (arm-lifting and spiking) after a 4-week training program than CT group.

The investigators plan to recruit 50 volleyball athletes. The sample size will be determined by previous studies and our future pilot study. It will be based on a significance level of 0.05, and a power of 0.80 to detect a difference on scapular upward rotation of 4° with a standard deviation of 4.5°. Based on these criteria, at least 21 participants with secondary shoulder impingement syndrome will be required in each group. To account for a withdrawal rate of 10%, participants will be included at least in each group. They will mainly be recruited from the universities in Taipei. A physical therapist will first evaluate the subject whether they are diagnosed of scapular dyskinesia. For subjects' evaluation, physical examination will include observation, palpation, selective tissue tension test (STTT), impingement sign test (Neer's, Hawkins-Kennedy), and scapular motor control test (flexion, abduction, external/internal rotation). Moreover, the investigators will design a check list to confirm whether they meet the inclusion/exclusion criteria. Patients who meet the criteria will enroll in this study, and then each of them will randomly be divided into two training groups.

The self-reported worst pain in the previous week will be measured using the visual analog scale (VAS; maximum score = 10 cm). The VAS is a self-reporting tool used to assess the level of pain of patients with shoulder pain due to scapular dyskinesis. Patients will be asked to draw a mark along a 10-cm line that indicates the amount of pain they are experiencing relative to a score of 0, indicating no pain, and a score of 10, indicating the most pain (worst). On the VAS, the investigators will choose to measure the "worst" pain, because previous studies suggested that it was more reliable than measuring "usual" pain.

LIBERTY™ electromagnetic tracking system (Polhemus, Colchester, VT, USA) was used to collect three-dimensional kinematic (3D) data during arm-lifting task and spiking task at a sampling rate of 120 Hz, and the software Motion Monitor® (Innovative Sport Training, Inc., Chicago. IL. USA) was used to analyze the data. The main measurement of shoulder kinematics include scapular upward/downward rotation, internal/external rotation, and anterior/posterior tilting. A stylus was used to digitize the bony landmarks for defining the anatomical coordinate system. The methods for this measure have been described previously.

For collecting muscle activation data, the investigators used surface electromyography (sEMG, TeleMyo 2400 G2 Telemetry; Noraxon USA, Inc., USA) to collect scapular muscles' activation during arm-lifting task. The investigators will measure the muscle activities of SA, UT, and LT. The electrodes will be placed according to previous studies, and will be positioned in parallel to the direction of the muscle ﬁbers.

For exercise performance assessment during spiking task, the investigators measured scapular kinematics consistency. The spiking task is consisted of total 30 rep of spiking, including initial 5 trials, 20 rep of fatigue, and last 5 trials. The investigators will conduct a pilot study to confirm the measurement which the investigators designed with enough reliability and validity.

The data of each outcome measures would collect at before (PRE measurement) and after 4-week intervention (POST measurement) except for self-reported pain (VAS), which would be collected at each end of week in addition. If the subject could not complete PRE and/or POST measurement, the investigators will note the reason which makes him/her unable to finish the whole trials, such as pain, instability or any discomfort.

Statistical analysis will be done on intention-to-treat basis using SPSS software (version 20; formerly SPSS Inc, now IBM Corporation, Armonk, NY). Missing data will be replaced using a conservative method with the last score carried forward. The independent t test or Chi-square test will be used for baseline demographic data. Descriptive statistics will include mean, standard deviation, and 95% confidence interval values, and the investigators will calculate 2 × 2 analyses of variance (ANOVAs; group × time; p < 0.05) for each outcome variables. Signiﬁcant differences revealed by the ANOVA will be further examined using Bonferroni post hoc analysis. The alpha (α) level will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Volleyball athletes who performed related sport activities for more than 10 hour/wks
* Age 18-30 years, with diagnosed of scapula dyskinesia by a physical therapist
* Shoulder girdle passive range of motion (PROM) within normal limitation
* Visual analog score (VAS) rating of pain during activities of sport or daily living during the previous week at a minimum of 3 cm on a 10-cm scale
* Insidious onset of symptoms unrelated to trauma and persistent for at least 4 wks

Exclusion Criteria:

* Can't finish the data collection process due to any other current musculoskeletal pain/injuries
* Any neuromuscular disorder, joint or bone disease
* History of any orthopedic surgeries

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-11-25 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Scapular movement consistency (Proprioceptive Feedback Magnitude, PFM) | Baseline and 4-week intervention
  Scapular positioning (kinematics) during spiking task (spike for 30 repetition, and compare the average of first and last 3 trials)

SECONDARY OUTCOMES:
Scapulo-humeral rhythm (scapular kinematics) | Baseline and 4-week intervention
  Scapular kinematics during spiking task
Scapula motor control (muscle activation percentage) | Baseline and 4-week intervention
  Scapular muscles' activation during spiking task
Self-reported pain (Visual Analogue Scale, VAS) | Baseline, end of week 1 treatment, end of week 2 treatment, end of week 3 treatment, and end of week 4 treatment
  The self-reported worst pain in spiking during previous one week (on a 10-cm scale, 0 cm = no pain, 10 cm = the most severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Fen Shih, PhD, Study Director — Department of Physical Therapy and Assistive Technology, National Yang-Ming University
Locations (1):
- National Yang Ming University, Taipei, Taiwan

REFERENCES:
- [Derived] Chang CC, Chang CM, Shih YF. Kinetic Chain Exercise Intervention Improved Spiking Consistency and Kinematics in Volleyball Players With Scapular Dyskinesis. J Strength Cond Res. 2022 Oct 1;36(10):2844-2852. doi: 10.1519/JSC.0000000000003904. Epub 2020 Dec 9. PMID 33306587